CLINICAL TRIAL: NCT04860089
Title: The Impact of Medical Cannabis on Pain and Inflammation in People Living With HIV
Brief Title: Pain, Inflammation, and Cannabis in HIV
Acronym: PITCH-E
Status: Withdrawn | Type: Observational
Why Stopped: This protocol was never initiated. Due to a change in funding, a new study will be registered in its place.
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Colorado, Boulder (Other); University of Pittsburgh (Other); Vireo Health (Other)
Responsible Party: Principal Investigator, Deepika Slawek, Assistant Professor of Medicine, Montefiore Medical Center
Other Study IDs: 2019-10394; GRANT13267147 (Other Grant/Funding Number: NIDA); 1K23DA053997-01A1 (NIH)
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections; Neuropathic Pain; Cannabis
MeSH Terms: conditions — HIV Infections; Neuralgia; Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will examine how medical cannabis use affects neuropathic pain, inflammation and adverse events in people living with HIV (PLWH) with neuropathic pain. We will study how varying ratios of THC and CBD in medical cannabis impact neuropathic pain, inflammation and adverse events.

DETAILED DESCRIPTION:
This study will examine how medical cannabis use affects neuropathic pain in PLWH with neuropathic pain. We will enroll adults with HIV who have a) neuropathic pain, b) are actively certified for medical cannabis, and c) intend to have soft gel capsule products dispensed at Vireo (medical cannabis dispensary) (including a high THC:low CBD product, an equal THC:CBD product, and a low THC:high CBD product). Over 14 weeks, data sources will include questionnaires, blood samples, urine samples; medical, pharmacy, and Prescription Monitoring Program (PMP) records. The primary independent variable will be type of medical cannabis product dispensed at dispensary, and the primary outcome will be self-reported pain.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* Diagnosis of HIV
* Fluency in English
* Active certification for medical cannabis
* No medical cannabis dispensed or used within the previous 30 days
* Intends to purchase soft-gel capsule medical cannabis at Vireo
* ICD-10 diagnosis code for neuropathic pain, OR
* Neuropathic pain in problem list of electronic medical record, OR
* Neuropathic pain questionnaire-short form>0

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete 14 weeks of study visits
* Medical cannabis use within 30 days prior to enrollment
* Unique pain symptoms (e.g. multiple sclerosis, rheumatoid arthritis)
* Terminal illness
* Current or prior psychotic disorder
* Street cannabis, opioid, cocaine, or benzodiazepine use in the past 30 days
* Dispensed opioids of benzodiazepines within 60 days
* Non-steroidal anti-inflammatory use within 7 days prior to enrollment
* Steroid use within the past 14 days with duration of therapy >=21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with HIV and neuropathic pain, who are not taking opioids and are actively certified for medical cannabis in New York
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-12-12 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain severity | 14 weeks
  self-reported pain severity measured via the Brief Pain Interference (BPI) severity scale (1-10) with higher score indicating worse pain. Measured weekly with web- or phone-based questionnaire.

SECONDARY OUTCOMES:
Circulating levels of inflammatory cytokines | 14 weeks
  Tests levels of recent inflammation (panel of inflammatory markers) at two time points before starting medical cannabis and 14 weeks after starting medical cannabis. Reported in pg/mL
Antiretroviral adherence | 14 weeks
  Measured at 0 and 14 weeks Visual Analog Scale [VAS] (0-100) with higher number indicating better adherence.
HIV Viral load suppression | 14 weeks
  HIV viral load measured at two time points (baseline and 14 weeks; copies/mL)
Depression | 14 weeks
  Measured at 0 and 14 weeks with the Patient Health Questionnaire- 9 [PHQ-9] (0-27) with higher score indicating worse depression
Anxiety | 14 weeks
  Measured at 0 and 14 weeks with the Generalized Anxiety Disorder-7 [GAD-7] (0-21) with higher score indicating worse anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Deepika E Slawek, MD, MPH, MS, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No